CLINICAL TRIAL: NCT00459628
Title: Randomized Trial Comparing Conventional vs Short-course Reduced Volume Conformal Post-surgery Radiation Treatment in Women With Stage I or II Breast Cancer
Brief Title: Trial of Tomotherapy in Breast Cancer
Acronym: TomoBreast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Vincent Vinh-Hung, MD, PhD, Clinical Professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007/009; 2007-002025-69 (EudraCT Number); SCIE2006-30 (Other Grant/Funding Number: Stichting tegen Kanker); ANI47 (Other: VUB)
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Breast Neoplasms
Keywords: early breast cancer; post-operative radiation treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional radiotherapy (Active Comparator): Conventional Long schedule Radiotherapy Arm
  Interventions: Radiation: Conventional radiotherapy
- Tomotherapy (Experimental): Short course schedule by tomotherapy
  Interventions: Radiation: Tomotherapy

INTERVENTIONS:
Radiation: Conventional radiotherapy — Radiation treatment delivered by conventional linear accelerator using matching fields
  Other Names: Arm I, Long schedule
  Arms: Conventional radiotherapy
Radiation: Tomotherapy — CT image guided intensity modulated radiation therapy delivered by the Tomotherapy HiArt system
  Other Names: Arm II, Short schedule, Helical Tomotherapy
  Arms: Tomotherapy

SUMMARY:
Tomotherapy is a new radiation therapy system that uses an integrated CT scanner during delivery of radiation treatment to improve the accuracy of the treatment. Furthermore the irradiation is delivered helicoidally allowing highly conformal shaping of dose distribution. However the magnitude of the clinical advantage of using the system in breast cancer is unknown. The purpose of the present study is to investigate whether or not the Tomotherapy can substantially reduce pulmonary and cardiac toxicities, as compared with conventional radiotherapy.

DETAILED DESCRIPTION:
Prior to surgery: histological confirmation; medical imaging.

Localizing markers are placed in case of breast conserving surgery.

After surgery, patients are randomized to one of two treatment arms:

* Arm I: radiotherapy using tangential chest fields, and supraclavicular field in case of nodal involvement, according to our hospital's standard procedure (Voordeckers M et al, Radiother Oncol 2003;68:227 and 2004;70:225). Dose-fractionation: 50 Gy in 25 fractions over 5 weeks, 2 Gy/fraction. Additional boost 16 Gy in 8 fractions over 2 weeks if breast conserving surgery (verify marker/clip localization) and age <= 70 years.
* Arm II: radiotherapy using the Tomotherapy system. Target area (breast, thorax wall, nodal areas) delimited according to pre-operative imaging and pathological description. Dose-fractionation (adapted from Whelan T et al, JNCI 2002;94:1143): 42 Gy in 15 fractions over 3 weeks, 2.8 Gy/fraction. Simultaneous boost 0.6 Gy/fraction if breast conserving surgery.

Physics quality control is integrated during treatment in both arms.

Radiotherapy begins within 6 weeks after the last breast surgery. Concurrent or sequential adjuvant systemic treatments are allowed. In case of sequential adjuvant treatment with chemotherapy first, radiotherapy begins within 6 weeks after completion of the adjuvant chemotherapy.

Quality of life, arm mobility and edema, pulmonary and heart function are assessed prior to radiotherapy, at 1-3 months after completion of radiotherapy, then yearly.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histologically proven breast carcinoma
* Stage I or II (T1-3N0 or T1-2N1 M0, AJCC/TNM 6th edition)
* Surgery with clear margins
* Pre-operative medical imaging (at least CT, MRI, and/or PET-scan)

Exclusion Criteria:

* Prior breast or thoracic radiotherapy
* Pregnancy or lactation
* Fertile patients without effective contraception
* Psychiatric or addictive disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2007-05; Primary Completion 2011-08 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pulmonary function and heart function tests | From end of treatment up to 3 years after treatment
  Assessment by pulmonary function tests and by heart echocardiography, compared with test values prior to treatment

SECONDARY OUTCOMES:
Local-regional recurrences. | From end of treatment up to 15 years after treatment
  Local-regional recurrences are assessed at time intervals as per the institution's standard practice for the clinical surveillance of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mark De Ridder, MD, PhD, Study Director — Radiotherapy Department, Universitair Ziekenhuis Brussel; Vincent Vinh-Hung, MD, PhD, Principal Investigator — Radiotherapy-Oncology, Universitair Ziekenhuis Brussel
Locations (1):
- Oncologisch Centrum, UZ Brussel, Jette, Brussels Capital, Belgium

REFERENCES:
- [Background] Voordeckers M, Van de Steene J, Vinh-Hung V, Storme G. Adjuvant radiotherapy after mastectomy for pT1-pT2 node negative (pN0) breast cancer: is it worth the effort? Radiother Oncol. 2003 Sep;68(3):227-31. doi: 10.1016/s0167-8140(03)00234-2. PMID 13129629
- [Background] Voordeckers M, Vinh-Hung V, Van de Steene J, Lamote J, Storme G. The lymph node ratio as prognostic factor in node-positive breast cancer. Radiother Oncol. 2004 Mar;70(3):225-30. doi: 10.1016/j.radonc.2003.10.015. PMID 15064006
- [Background] Whelan T, MacKenzie R, Julian J, Levine M, Shelley W, Grimard L, Lada B, Lukka H, Perera F, Fyles A, Laukkanen E, Gulavita S, Benk V, Szechtman B. Randomized trial of breast irradiation schedules after lumpectomy for women with lymph node-negative breast cancer. J Natl Cancer Inst. 2002 Aug 7;94(15):1143-50. doi: 10.1093/jnci/94.15.1143. PMID 12165639
- [Result] Versmessen H, Vinh-Hung V, Van Parijs H, Miedema G, Voordeckers M, Adriaenssens N, Storme G, De Ridder M. Health-related quality of life in survivors of stage I-II breast cancer: randomized trial of post-operative conventional radiotherapy and hypofractionated tomotherapy. BMC Cancer. 2012 Oct 25;12:495. doi: 10.1186/1471-2407-12-495. PMID 23098579
- [Result] Van Parijs H, Miedema G, Vinh-Hung V, Verbanck S, Adriaenssens N, Kerkhove D, Reynders T, Schuermans D, Leysen K, Hanon S, Van Camp G, Vincken W, Storme G, Verellen D, De Ridder M. Short course radiotherapy with simultaneous integrated boost for stage I-II breast cancer, early toxicities of a randomized clinical trial. Radiat Oncol. 2012 Jun 1;7:80. doi: 10.1186/1748-717X-7-80. PMID 22656865
- [Result] Adriaenssens N, De Ridder M, Lievens P, Van Parijs H, Vanhoeij M, Miedema G, Voordeckers M, Versmessen H, Storme G, Lamote J, Pauwels S, Vinh-Hung V. Scapula alata in early breast cancer patients enrolled in a randomized clinical trial of post-surgery short-course image-guided radiotherapy. World J Surg Oncol. 2012 May 16;10:86. doi: 10.1186/1477-7819-10-86. PMID 22591589
- [Result] Adriaenssens N, Vinh-Hung V, Miedema G, Versmessen H, Lamote J, Vanhoeij M, Lievens P, van Parijs H, Storme G, Voordeckers M, De Ridder M. Early contralateral shoulder-arm morbidity in breast cancer patients enrolled in a randomized trial of post-surgery radiation therapy. Breast Cancer (Auckl). 2012;6:79-93. doi: 10.4137/BCBCR.S9362. Epub 2012 Jul 30. PMID 22904635
- [Result] Verbanck S, Hanon S, Schuermans D, Van Parijs H, Vinh-Hung V, Miedema G, Verellen D, Storme G, Vanhoeij M, Lamote J, De Ridder M, Vincken W. Small airways function in breast cancer patients before and after radiotherapy. Breast Cancer Res Treat. 2012 Oct;135(3):857-65. doi: 10.1007/s10549-012-2201-7. Epub 2012 Aug 22. PMID 22910929
- [Derived] Van Parijs H, Cecilia-Joseph E, Gorobets O, Storme G, Adriaenssens N, Heyndrickx B, Verschraegen C, Nguyen NP, De Ridder M, Vinh-Hung V. Lung-heart toxicity in a randomized clinical trial of hypofractionated image guided radiation therapy for breast cancer. Front Oncol. 2023 Nov 20;13:1211544. doi: 10.3389/fonc.2023.1211544. eCollection 2023. PMID 38053657
- [Derived] Van Parijs H, Vinh-Hung V, Fontaine C, Storme G, Verschraegen C, Nguyen DM, Adriaenssens N, Nguyen NP, Gorobets O, De Ridder M. Cardiopulmonary-related patient-reported outcomes in a randomized clinical trial of radiation therapy for breast cancer. BMC Cancer. 2021 Nov 4;21(1):1177. doi: 10.1186/s12885-021-08916-z. PMID 34736429